CLINICAL TRIAL: NCT05688293
Title: Gingival Recession (RT1) Treatment With Different Gingival Augmentation Surgeries Compared With Untreated Contralateral Sites: A Randomized Controlled Clinical Study
Brief Title: Gingival Recession (RT1) Treatment With Different Gingival Augmentation Surgeries
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Misr International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PER 5213005
Record Dates: First submitted 2023-01-06; First posted 2023-01-18 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-01

CONDITIONS: Gingival Recession
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Intervention Model Description: Three parallel groups
Who Masked: Participant, Outcomes Assessor
Masking Description: the patient won't know the type of the procedures done to him The outcome assessor won't know which group he the is assessing it's results
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Connective tissue graft (Active Comparator): Patients will receive non-surgical periodontal treatment and connective tissue graft using tunneling technique
  Interventions: Procedure: Connective tissue graft
- Free gingival Graft (Active Comparator): Patients will receive non-surgical periodontal treatment and partially de-epithelized free gingival graft
  Interventions: Procedure: Free gingival graft
- Non surgical procedure (Active Comparator): Patients will receive non-surgical periodontal treatment only
  Interventions: Procedure: Non surgical

INTERVENTIONS:
Procedure: Connective tissue graft — non-surgical periodontal treatment and connective tissue graft
  Arms: Connective tissue graft
Procedure: Free gingival graft — will receive non-surgical periodontal treatment and partially de-epithelized free gingival graft
  Arms: Free gingival Graft
Procedure: Non surgical — non-surgical periodontal treatment only
  Arms: Non surgical procedure

SUMMARY:
Thin gingival phenotype is one of the major causative factors of gingival recession type 1 which can result in hypersensitivity, discomfort, and compromised esthetics. This study assess the efficacy of increasing the gingival thickness from thin gingival phenotype to thick gingival phenotype in the treatment of patients suffering from gingival recession (RT1) and maintenance of results using either connective tissue graft or de-epithelized free gingival graft after non-surgical periodontal debridement compared to non-surgical periodontal debridement alone.

DETAILED DESCRIPTION:
This parallel arm randomized controlled clinical trial study will include systematically free patients with thin gingival phenotype. They will be randomly allocated to three equal groups. Group A (test group, n=10) will receive non-surgical periodontal treatment and connective tissue graft using tunneling technique, Group B (test group, n=10) will receive non-surgical periodontal treatment and partially de-epithelized free gingival graft, while group C (control group, n=10) will receive non-surgical periodontal treatment only. After 3, 6 and 12 months gingival biotype will be clinically assessed (1ry outcome). This parameter will be recorded at baseline, 3, 6 and 12 months. The 2ry outcomes will include recording of recession depth, plaque index, bleeding on probing, keratinized tissue width . Postoperative pain and swelling will be recorded daily by the patient for the 1st two weeks post-surgically. Postoperative instructions and medication will be given to the patient. All readings will be carried out by a calibrated outcome assessor who will be masked. Follow-up will be performed to assess the outcomes and to ensure performing proper oral hygiene. Data collected will be tabulated and statistically analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Medically free patients (American Society of Anesthesiologists I; ASA I)
* Patients diagnosed with recession (RT1)
* Fair oral hygiene
* Patient accepting to provides an informed consent and the follow-up

Exclusion Criteria:

* Carious teeth and teeth with periapical infection.
* Patients diagnosed with periodontitis
* Smokers
* Pregnant and lactating females

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-02-05 (Actual); Primary Completion 2026-01-20 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Gingival phenotype change | at baseline 3,6 and 12 months
  determination of the change in gingival thickness in mm using periodontal probe

SECONDARY OUTCOMES:
Keratinized tissue width | at baseline 3,6 and 12 months
  determination of Keratinized tissue width in mm using periodontal probe
Root coverage esthetic score (RES) | at baseline 3,6 and 12 months
  It is a scoring system to assess the level of gingival margin (GM),marginal tissue contour (MTC),Soft tissue texture, Mucogingival alignment (MGJ),Gingival color The score is 0,1 and 3 where 0 is the minimum and 3 is the maximum

CONTACTS AND LOCATIONS:
Overall Officials: Zainab Hafez, Lecturer, Principal Investigator — Lecturer, faculty of oral and dental medicine misr international university; Shahinaz Al ashiry, Asso. Prof, Study Director — Associate professor, faculty of oral and dental medicine misr international university; Yahia Amer, Lecturer, Principal Investigator — Lecturer, faculty of oral and dental medicine misr international universit
Locations (1):
- Faculty of oral and dental medicine, Misr international university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No